CLINICAL TRIAL: NCT03943849
Title: The Use of Dental Pulp Tissue as an Autogenous Graft for Ridge Augmentation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Karo Parsegian, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-DB-18-0873
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Tooth Loss
Keywords: Bone graft; Tooth extraction; Dental pulp
MeSH Terms: conditions — Tooth Loss | interventions — Sutures

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Particulate bone graft plus autogenous dental pulp tissue (Experimental): Dental pulp will be isolated from teeth extracted for non-periodontal reasons chairside. The isolated dental pulp will be mixed with hydrated particulate bone graft, and the mixture will be placed in the debrided extraction socket. The socket will be covered by a resorbable collagen membrane and sutured.
  Interventions: Other: Particulate bone graft; Other: Autogenous dental pulp tissue; Other: Resorbable collagen membrane; Other: Suture
- Particulate bone graft (Active Comparator): Hydrated particulate bone graft will be placed in the debrided extraction socket. The socket will be covered by a resorbable collagen membrane and sutured.
  Interventions: Other: Particulate bone graft; Other: Resorbable collagen membrane; Other: Suture

INTERVENTIONS:
Other: Particulate bone graft — Creos allo.gain allogenic bone particulate mineralized cortical bone will be hydrated and placed in the extraction socket.
  Other Names: creos allo.gain; allogenic bone particulates
Other: Autogenous dental pulp tissue — Dental pulp will be isolated from teeth extracted for non-periodontal reasons chairside, mixed with hydrated particulate bone graft, and then placed in the extraction socket.
  Arms: Particulate bone graft plus autogenous dental pulp tissue
Other: Resorbable collagen membrane — After placement of particulate bone graft or particulate bone graft plus autogenous dental pulp tissue, socket will be covered by a resorbable collagen membrane and sutured.
Other: Suture — Resorbable or non-resorbable suture material

SUMMARY:
The purpose of this study is to examine and compare the effects of autogenous dental pulp tissue on bone formation in the extraction sockets as compared to commonly used particulate bone graft. The effects on bone formation will be examined using a wide variety of assays.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Physical Status Classification System ASA 1 (A normal healthy patient) or ASA 2 (A patient with mild systemic disease)
* never smoker
* patients with planned tooth extraction
* intact extraction sockets
* no medication or antibiotics intake for at least 6 months prior to the procedure
* patients who gave their consent to participate in the study.

Exclusion Criteria:

* vulnerable subjects (children, pregnant and lactating women, patients with learning disabilities, and prisoners)
* inability to obtain pulp tissue (for example, due to previous endodontic therapy, obliterated pulp canals)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Bone fill as assessed by radiograph | immediately after placement of bone graft
Bone fill as assessed by radiograph | 2 months after placement of bone graft
Bone fill as assessed by radiograph | 4 months after placement of bone graft

SECONDARY OUTCOMES:
Extent of mineralization as assessed by von Kossa staining | 4 months after placement of bone graft
Extent of mineralization as assessed by Xylenol Orange staining | 4 months after placement of bone graft
Expression of osteoblastic marker Bsp assessed by quantitative PCR (qPCR) | 4 months after placement of bone graft
Expression of osteoblastic marker BSP assessed by immunostaining using anti-BSP antibody | 4 months after placement of bone graft
Expression of osteoblastic marker Bglap assessed by quantitative PCR (qPCR) | 4 months after placement of bone graft
Expression of osteoblastic marker BGLAP assessed by immunostaining using anti-BGLAP antibody | 4 months after placement of bone graft
Expression of osteoblastic marker Dmp1 assessed by quantitative PCR (qPCR) | 4 months after placement of bone graft
Expression of osteoblastic marker DMP1 assessed by immunostaining using anti-DMP1 antibody | 4 months after placement of bone graft
Expression of osteoblastic marker Col1a1 assessed by quantitative PCR (qPCR) | 4 months after placement of bone graft
Expression of osteoblastic marker Sost assessed by quantitative PCR (qPCR) | 4 months after placement of bone graft

CONTACTS AND LOCATIONS:
Overall Officials: Karo Parsegian, DMD, MDSc, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No